CLINICAL TRIAL: NCT07251023
Title: Multicenter Randomized Double-blind Placebo-controlled Active Comparator-controlled Study to Assess the Efficacy and Safety of DMB-I (Dimebon®, INN: Latrepirdine) in Patients With Dementia Associated With Alzheimer's Disease
Brief Title: Efficacy and Safety of DMB-I (INN: Latrepirdine) in Patients With Alzheimer Type Dementia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bigespas LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMBN_ALZH-2025-III
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Type Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine; Memantine

STUDY DESIGN:
Intervention Model Description: placebo-controlled and active comparator-controlled two-stage study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DMB-I (INN: Latrepirdine) (Experimental): DMB-I (INN: Latrepirdine), 10 mg, 2 tablets 3 times daily (Group 3: DMB-I)
  Interventions: Drug: DMB-I (INN: Latrepirdine)
- Placebo + Memantine Hydrochloride (Placebo Comparator): Placebo, 2 tablets 3 times daily + Akatinol Memantine®, 20 mg once daily (Group 2: Placebo + Memantine).
  Interventions: Drug: Memantine Hydrochloride 20 MG; Drug: Placebo
- DMB-I (INN: Latrepirdine) + Memantine Hydrochloride (Active Comparator): DMB-I (INN: Latrepirdine), 10 mg, 2 tablets 3 times daily + Akatinol Memantine®, 20 mg once daily (Group 1: DMB-I + Memantine)
  Interventions: Drug: DMB-I (INN: Latrepirdine); Drug: Memantine Hydrochloride 20 MG

INTERVENTIONS:
Drug: DMB-I (INN: Latrepirdine) — Active agent: Dimethylmethylpyridinylethyltetrahydrocarboline. Investigational drug in the study
  Other Names: Latrepirdine, Dimebon®
  Arms: DMB-I (INN: Latrepirdine); DMB-I (INN: Latrepirdine) + Memantine Hydrochloride
Drug: Memantine Hydrochloride 20 MG — Memantine is used to treat moderate to severe Alzheimer's disease. Active comparator drug in the study
  Other Names: Akatinol Memantine®
  Arms: DMB-I (INN: Latrepirdine) + Memantine Hydrochloride; Placebo + Memantine Hydrochloride
Drug: Placebo — Placebo comparator (dummy) in the study.
  Arms: Placebo + Memantine Hydrochloride

SUMMARY:
The goal of this clinical study is to learn if the study drug DMB-I (INN: Latrepirdine) works to treat Alzheimer type dementia in adults. It will also learn about the safety of DMB-I (INN: Latrepirdine).

The main questions it aims to answer are:

* Does DMB-I improve cognitive functions in patients with dementia associated with Alzheimer's disease, and how sigificant the improvement is?
* What medical problems do participants have when taking DMB-I? Researchers will compare DMB-I to a placebo (a look-alike substance that contains no drug) to see if the study drug works to treat Alzheimer type dementia.
* Is DMB-I effective and safe when taken long-term?

Participants will:

Take the study drug or a placebo (with or without Akatinol Memantine®) every day for 26 weeks at Stage 1 of the study, and take the study drug (with or without Akatinol Memantine®) every day for 26 weeks at Stage 2 of the study.

Visit the clinic 13 times for checkups and tests Keep a diary of their symptoms

DETAILED DESCRIPTION:
This is a multicenter randomized double-blind placebo-controlled two-stage study that is to assess efficacy and safety of DMB-I (INN: Latrepirdine) in patients with Alzheimer type dementia.

The study is planned to be conducted in approximately 15 clinical sites of the Russian Federation.

At Stage 1 (comparative stage, 26 weeks), the study will examine three treatment groups. Patients in Group 1 and Group 2 will receive Akatinol Memantine® in addition to the study therapy (DMB-I or Placebo). Patients in Group 3 will receive DMB-I alone. The study is double-blind for DMB-I and Placebo; Akatinol Memantine® will not be blinded.

Patients meeting all the eligibility criteria will be randomized into one of three treatment groups:

1. DMB-I, 10 mg, 2 tablets 3 times daily + Akatinol Memantine®, 20 mg once daily - 175 patients (Group 1: DMB-I + Memantine).
2. Placebo, 2 tablets 3 times daily + Akatinol Memantine®, 20 mg once daily - 175 patients (Group 2: Placebo + Memantine).
3. DMB-I, 10 mg, 2 tablets 3 times daily - 100 patients (Group 3: DMB-I). Following completion of Stage 1, patients will continue participating in the open-label stage of the study (Stage 2) for additional 26 weeks to evaluate the long-term efficacy and safety of DMB-I. During this stage, patients in Group 1 (DMB-I + Memantine) will continue their study therapy unchanged. Patients in Group 2 (Placebo + Memantine) will discontinue Placebo and begin therapy with DMB-I (while continuing to take Akatinol Memantine®). Patients in Group 3 (DMB-I monotherapy) will also continue their therapy unchanged.

The total study duration for each patient is approximately 56 weeks broken down as follows:

Screening period: up to 2 weeks, Treatment period (Stage 1): 26 weeks, Treatment period (Stage 2): 26 weeks, Follow-up period: 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (Group 1 and Group 2):

  1. Informed consent to participate in the study.
  2. Patients of any gender aged 60 to 90 years inclusive.
  3. Patients diagnosed with mild to moderate Alzheimer type dementia according to the NINCDS-ADRDA criteria, receiving basic treatment with memantine at a daily dose of 20 mg for at least 2 months.
  4. The MMSE score is in the range of 10-23 inclusive.
  5. The ADAS-Cog score is in the range of 20-54 inclusive.
  6. No signs of dementia of vascular origin according to CT/MRI data. Repeated Acute Cerebrovascular Accidents (focal infarctions) in brain areas that are critical for cognitive functions and behavior are the mandatory neuroimaging signs of vascular dementia.
  7. The Modified Hachinski Ischemic Scale (HIS) score is < 7.
  8. The presence of a caregiver who is in contact with the patient a significant part of the time, agrees to accompany the patient to all visits, monitor the intake of the study drug and fill out the patient's diary.
  9. An ability to comply with all Protocol requirements.
* Inclusion Criteria (Group 3):

  1. Informed consent to participate in the study.
  2. Patients of any gender aged 60 to 90 years inclusive.
  3. Patients diagnosed with mild to moderate Alzheimer type dementia according to the NINCDS-ADRDA criteria, who are not receiving dementia-contolling medications (memantine, donepezil, rivastigmine, or galantamine) at screening or for the last two (or more) months prior to screening; however, taking such medications for more than two months prior to screening does not limit a patient's participation in the study.
  4. The MMSE score is in the range of 10-23 inclusive.
  5. The ADAS-Cog score is in the range of 20-54 inclusive.
  6. No signs of dementia of vascular origin according to CT/MRI data. Repeated Acute Cerebrovascular Accidents (focal infarctions) in brain areas that are critical for cognitive functions and behavior are the mandatory neuroimaging signs of vascular dementia.
  7. The Modified Hachinski Ischemic Scale (HIS) score is < 7.
  8. The presence of a caregiver who is in contact with the patient a significant part of the time, agrees to accompany the patient to all visits, monitor the intake of the study drug and fill out the patient's diary.
  9. An ability to comply with all Protocol requirements.

Exclusion Criteria:

1. Patients diagnosed with other diseases that cause dementia (severe hypothyroidism, anemia, brain tumor, neuroinfections, etc.) at screening.
2. History of other neurodegenerative diseases of the brain, Parkinson's disease, multiple sclerosis, demyelinating diseases of the nervous system, hereditary degenerative diseases of the central nervous system, abnormalities of the nervous system, uncontrolled epilepsy, hallucinations, other neurological disorders seriously affecting motor or cognitive function, in the opinion of the investigator.
3. History of intolerance to any of the components of the study drug.
4. History of stroke.
5. Active oncological process.
6. The need for surgeries on the vessels of the neck or brain, including endovascular interventions, during the study.
7. Signs of significant uncontrolled concomitant disease that, in the opinion of the Investigator, could prevent the patient from participating in the study, including:

   * Respiratory system disorders;
   * Cardiovascular system disorders;
   * Severe renal impairment (glomerular filtration rate <30ml/min);
   * Severe liver dysfunction (ALT, AST > 2 times the upper limit of normal);
   * Endocrine system disorders;
   * Gastrointestinal disorders.
8. Systemic autoimmune diseases or vascular collagenoses requiring previous or current treatment with systemic drugs.
9. Myocardial infarction within 12 months prior to screening.
10. Known systemic infection (viral hepatitis, HIV, tuberculosis, syphilis).
11. Life expectancy less than a year after randomization.
12. Use of drugs that negatively affect cognitive function (tricyclic antidepressants, benzodiazepines, antipsychotics, hypnotics, etc.), as well as drugs of prohibited therapy (including Cerebrolysin, preparations of ginkgo biloba extract, any other drugs with nootropic, antioxidant, metabolic effects, as well as drugs used to treat dementia) within 1 month prior to screening.
13. Moderate to severe depression (Hamilton scale score of 18 or more).
14. Smoking.
15. Episodes of alcohol or drug abuse within the last 6 months.
16. Inability to comply with study procedures even with the assistance, in the opinion of the investigator.
17. Participation in another clinical trial within the last 6 months.
18. Episodes of other serious or unstable psychiatric conditions that make the patient unsuitable for participation in a clinical study, alter the validity of obtaining an informed consent, or may affect the patient's ability to participate in the trial.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in ADAS-Cog Scale overall score at Week 26 compared to baseline (Week 0) in patients receiving DMB-I (Group 1) Vs. patients receiving placebo (Group 2) | Baseline (Week 0) Vs. Week 26
  ADAS-Cog Scale consists of 12 questions. The scale's minimum score - 0, maximum score - 88, where the higher score means the worse outcome

SECONDARY OUTCOMES:
Assessment of the change in ADAS-Cog Scale overall score at Week 26 compared to baseline (Week 0) in patients receiving DMB-I (Group 3) Vs. patients receiving placebo (Group 2) | Baseline (Week 0) Vs. Week 26
  ADAS-Cog Scale consists of 12 questions. The scale's minimum score - 0, maximum score - 88, where the higher score means the worse outcome
Change in ADAS-Cog Scale overall score at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  ADAS-Cog Scale consists of 12 questions. The scale's minimum score - 0, maximum score - 88, where the higher score means the worse outcome

OTHER OUTCOMES:
Change in ADAS-Cog component scores (Item 1: Word Learning, Item 4: Delayed Word Recall, Item 6: Ideational Praxis, Item 7: Orientation) at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  ADAS-Cog Scale consists of 12 questions. The scale's minimum score - 0, maximum score - 88, where the higher score means the worse outcome
Change in the Neuropsychiatric Inventory (NPI) behavioral symptom frequency and severity at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  The total NPI score is the sum of all individual domain scores, with a possible range of 0 to 144. A higher NPI total score indicates a greater number and more severe neuropsychiatric symptoms.
Change in Instrumental Activities of Daily Living (IADL) overall score at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  The scale is scored from 0 to 8, where a score of 8 indicates full independence and a score of 0 indicates complete dependence. The total score is calculated by summing the scores for each of the eight activities.
Change in Clinical Global Impression-Score (CGI-S) at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  This is a 7-point scale that rates the severity of a patient's illness based on a clinician's professional judgment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients), with 4 being "moderately ill".
Change in Clinical Global Impression-I (CGI-I) at Week 4, Week 12, Week 26, Week 30, Week 38, and Week 52 compared to baseline (Week 0) across all treatment groups | Baseline (Week 0) Vs. Week 4, Week 12, Week 26, Week 30, Week 38, Week 52
  This is a 7-point scale that rates the severity of a patient's illness based on a clinician's professional judgment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients), with 4 being "moderately ill".

CONTACTS AND LOCATIONS:
Locations (12):
- Russia (12):
  - State autonomous healthcare institution "Transregional Clinical Diagnostic Center", Kazan'
  - Moscow State budgetary healthcare institution "City Clinical Hospital named after V.M. Buyanov of the Moscow Healthcare Department", Moscow
  - Federal State Budgetary Institution "Federal Center for Brain and Neurotechnology" of the Federal Medical and Biological Agency, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Nizhny Novgorod region State budgetary healthcare institution " Nizhny Novgorod Clinical Psychiatric Hospital No. 1", Nizhny Novgorod
  - State budgetary healthcare institution "Leningrad Regional Mental Health Center", Roshchino
  - "Medical Center Nova Vita" LLC, Rostov-on-Don
  - Saint Petersburg State budgetary healthcare institution "Psychiatric Hospital No. 1 named after P.P. Kashchenko", Saint Petersburg
  - "Medical services" LLC, Saint Petersburg
  - Saint Petersburg State budgetary healthcare institution "Psychoneurologic dispensary № 5", Saint Petersburg
  - "Sphera Med" LLC, Saint Petersburg
  - Saint Petersburg State budgetary healthcare institution "City Hospital No. 40 of Kurortniy district", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No